CLINICAL TRIAL: NCT04986436
Title: A Phase I, Randomized, Double-blinded, Placebo-controlled Dose Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral Administered HS-10360 in Healthy Subjects.
Brief Title: Phase I Study to Evaluate Safety, Tolerability, and Pharmacokinetics of HS-10360 in Healthy Subjects.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10360-101
Record Dates: First submitted 2021-07-06; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: HS-10360; Safety; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10360 (Experimental): Either single or multiple doses of varying dose levels
  Interventions: Drug: HS-10360
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-10360 — Single or multiple dose(s) of HS-10360
  Arms: HS-10360
Drug: Placebo — Single or multiple dose(s) of Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of single and multiple oral administered doses of HS-10360 in healthy subjects.

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blinded, placebo-controlled, single ascending doses (SAD) study followed by multiple ascending doses (MAD) clinical trial to assess the safety, tolerability, and pharmacokinetics of HS-10360 tablet (s) in Chinese healthy adult subjects.

Approximately five sequential dose levels will be evaluated in SAD phase. Two sentinel subjects will be enrolled in the first cohort and minimal 72 hours post-dose safety data will be evaluated before the remaining subjects are enrolled in this cohort. Approximately three sequential dose cohorts (the specific dose levels should be further determined according to the SAD results) will be evaluated in MAD phase. Each subject will receive only one dose regimen in this study. Safety data up to Day12 (±2) in SAD and up to Day28 (±2) in MAD will be reviewed prior to the next dose level. The number of Cohorts in SAD and MAD would be adjusted based on the assessment of SRC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:
* Healthy male or female subjects between 18 and 45 years old;
* Body weight more than 50.0kg (male) or 45.0kg (female), body mass index (BMI) within the range of 19.0~26.0kg/m2 (both inclusive);
* Subjects and their partners should have no fertility plan, no sperm or ootid donation plan and must use highly effective contraceptive methods (such as abstinence, condom, etc.) from the screening period to 6 months post-trial;
* Additional inclusion criteria apply;

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Clinically significant abnormalities in baseline results of laboratory evaluations;
* Subjects has a positive result of any of following virology tests (hepatitis B surface antigen HBsAg, hepatitis B core antibody HBcAb, hepatitis C virus HCV antibody, human immunodeficiency virus HIV antibody, Treponema pallidum antibody TP-Ab) ;
* History or evidence of clinically significant cardiovascular, pulmonary, endocrine, gastrointestinal, psychiatric, neurologic, hematological or metabolic diseases, especially those conditions that interfere with absorption, metabolism and/or excretion of the study drug, determined by the investigator;
* Any previous or current severe infection, such as cellulitis, pneumonia, sepsis etc., requiring hospitalization and/or intravenous antibiotic treatment, within 30 prior to the screening period;
* Have participated in clinical trials of other drugs or medical devices within 3 months or within 5 half-lives of other drugs before screening (if 5 half-lives exceed 3 months);
* History or presence of allergy, especially known allergy to investigational product components or other JAK inhibitors;
* Had taken any medication, including prescription, over-the-counter, herbal, dietary supplements, or vaccines, within the previous 2 weeks; or within the five half-lives of the aforementioned drugs prior to randomization;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAE) | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experience one or more treatment-emergent adverse events (TEAE)
Moderate or severe treatment-emergent adverse events (TEAE) | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experience one or more moderate or severe treatment-emergent adverse events (TEAE)
Serious treatment-emergent adverse events (TEAE) | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experience one or more serious treatment-emergent adverse events (TEAE)
Clinical laboratory measurements | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experienced a clinically significant clinical laboratory measurements
Electrocardiogram | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experienced a clinically significant electrocardiogram (ECG) result
Vital Signs | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experienced a clinically significant vital sign measurement

SECONDARY OUTCOMES:
SAD pharmacokinetic endpoints: | Day1-Day6
  The maximum plasma concentration (Cmax)
SAD pharmacokinetic endpoints: | Day1-Day6
  Time to Cmax (Tmax)
SAD pharmacokinetic endpoints: | Day1-Day6
  The area under the plasma concentration-time curve from time zero to the time of the last measurable concentration (AUC0-t)
SAD pharmacokinetic endpoints: | Day1-Day6
  The area under the plasma concentration-time curve from time zero xtrapolated to infinite time (AUC0-∞)
SAD pharmacokinetic endpoints: | Day1-Day6
  Terminal rate constant (λz)
SAD pharmacokinetic endpoints: | Day1-Day6
  Half life (t½)
SAD pharmacokinetic endpoints: | Day1-Day6
  Apparent clearance following oral administration (CL/F)
SAD pharmacokinetic endpoints: | Day1-Day6
  Apparent volume of distribution following oral administration (Vz/F)
SAD pharmacokinetic endpoints: | Day1-Day6
  Mean residence time (MRT)
SAD pharmacokinetic endpoints: | Day1-Day6(SAD)
  Amount excreted in urine (Aeu)
SAD pharmacokinetic endpoints: | Day1-Day6(SAD)
  Amount excreted in feces (Aef)
MAD pharmacokinetic endpoints: | Day1-Day19
  The maximum steady state drug concentration in plasma during dosing interval (Css,max)
MAD pharmacokinetic endpoints: | Day1-Day19
  The minimum steady state drug concentration in plasma during dosing interval (Css,min)
MAD pharmacokinetic endpoints: | Day1-Day19
  Average steady state drug concentration in plasma during dosing interval Css,av)
MAD pharmacokinetic endpoints: | Day1-Day19
  Time to Css, max (Tss,max)
MAD pharmacokinetic endpoints: | Day1-Day19
  The area under the plasma concentration-time curve over the dosing interval at steady state (AUCss)
MAD pharmacokinetic endpoints: | Day1-Day19
  The area under the plasma concentration-time curve from time zero to the time of the last measurable concentration at steady state(AUC0-t)
MAD pharmacokinetic endpoints: | Day1-Day19
  The area under the plasma concentration-time curve from time zero xtrapolated to infinite time (AUC0-∞) at steady state
MAD pharmacokinetic endpoints: | Day1-Day19
  Half life (t½)
MAD pharmacokinetic endpoints: | Day1-Day19
  Accumulation ratio (Rac)
MAD pharmacokinetic endpoints: | Day1-Day19
  Apparent clearance at steady state following oral administration (CLss/F)
MAD pharmacokinetic endpoints: | Day1-Day19
  Apparent volume of distribution at steady state following oral administration (Vd/F)
MAD pharmacokinetic endpoints: | Day1-Day19
  Amount excreted in urine (Aeu)
MAD pharmacokinetic endpoints: | Day1-Day19
  Amount excreted in feces (Aef)

CONTACTS AND LOCATIONS:
Overall Officials: Qing He, bachelor, Principal Investigator — Wu Xi people's hospital